CLINICAL TRIAL: NCT02060721
Title: MERIT-2 : Long Term, Multicenter, Single-arm, Open-label Extension Study of the MERIT-1 Study, to Assess the Safety, Tolerabilty and Efficacy of Macitentan in Subjects With Inoperable Chronic Thromboembolic Pulmonary Hypertension (CTEPH)
Brief Title: Clinical Study to Assess the Safety, Tolerability and Efficacy of Macitentan in Subjects With Inoperable Chronic Thromboembolic Pulmonary Hypertension
Acronym: MERIT-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-055E202; 2013-003457-25 (EudraCT Number)
Record Dates: First submitted 2014-01-02; First posted 2014-02-12 (Estimated); Results first posted 2023-04-11 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: Chronic thromboembolic pulmonary hypertension (CTEPH)
MeSH Terms: interventions — macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Macitentan (Experimental): Macitentan 10mg, oral tablet, once daily
  Interventions: Drug: Macitentan

INTERVENTIONS:
Drug: Macitentan — Macitentan 10mg, oral tablet, once daily
  Other Names: ACT-064992

SUMMARY:
Long-term study to evaluate if macitentan is safe, tolerable and efficient enough to be used for treatment of inoperable chronic thromboembolic pulmonary hypertension (CTEPH)

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Subject with CTEPH having completed the double-blind (DB) AC-055E201/ MERIT-1 study as scheduled (i.e., who remained in the DB study up to Week 24).
* Females of childbearing potential must have a negative pre-treatment serum pregnancy test, be advised on appropriate methods of contraception, and agree to use 2 reliable methods of contraception.

Exclusion Criteria:

* Permanent discontinuation of DB study treatment due to an hepatic adverse event or liver aminotransferase abnormalities.
* Any known factor (e.g., drug or substance abuse) or disease (e.g., unstable psychiatric illness) that, in the opinion of the investigator, may interfere with treatment compliance or interpretation of the results, or that may influence the ability to comply with any of the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin McGuire, Study Director — Actelion
Locations (33):
- Leuven, Belgium
- China (5):
  - Beijing
  - Guangzhou
  - Shanghai
  - Shenyang
  - Wuhan
- Prague, Czechia
- France (3):
  - Le Kremlin-Bicêtre
  - Paris
  - Toulouse
- Germany (3):
  - Giessen
  - Heidelberg
  - Würzburg
- Hungary (2):
  - Budapest
  - Debrecen
- Kaunas, Lithuania
- Mexico City, Mexico
- Poland (2):
  - Lublin
  - Wroclaw
- Russia (5):
  - Kemerovo
  - Moscow
  - Novosibirsk
  - Saint Petersburg
  - Tomsk
- Zurich, Switzerland
- Thailand (2):
  - Bangkok
  - Chiang Mai
- Capa_Istanbul, Turkey (Türkiye)
- Ukraine (2):
  - Kyiv
  - Lviv
- United Kingdom (3):
  - Cambridge
  - London
  - Sheffield

REFERENCES:
- [Derived] Kim NH, D'Armini AM, Howard LS, Jenkins DP, Jing ZC, Mayer E, Chamitava L, Lack G, Rofael H, Solonets M, Ghofrani HA. Long-Term Safety and Efficacy of Macitentan in Inoperable Chronic Thromboembolic Pulmonary Hypertension: Results from MERIT and its Open-Label Extension. Pulm Ther. 2025 Mar;11(1):101-116. doi: 10.1007/s41030-024-00276-w. Epub 2024 Nov 9. PMID 39520648

RESULTS

PARTICIPANT FLOW:
Groups:
- Macitentan 10 Milligrams (mg): Eligible participants who were either randomized to macitentan 10 mg or placebo group during 24 weeks double-blind MERIT-1 (NCT02021292) study, were rolled-over to this open-label extension study and received macitentan 10 mg tablet orally once daily starting from Day 1 to the end of treatment (treatment exposure ranged from 1 to 82 months).
Period: Overall Study
Arm/Group | Macitentan 10 Milligrams (mg)
Started | 76
Completed | 38
Not Completed | 38
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 2
Not completed — Death | 14
Not completed — Withdrawal by Subject | 2
Not completed — Compliance with local regulation: enrolled in China | 19

BASELINE CHARACTERISTICS:
Arm/Group | Macitentan 10 Milligrams (mg)
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (13.99) [lower limit 13.99]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 74
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 27
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 49
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study. TEAEs are those events that started after administration of the first dose and up to safety follow-up visit/end of study, that is, 30 days after the last dose of study medication.
Time Frame: Up to 30 days after study treatment discontinuation (treatment exposure ranged from 1 to 82 months)
Population: Open-label analysis set (OLAS) included all data from participants who were enrolled into this open-label extension study, from the time they entered this open-label extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 Milligrams (mg)
Number analyzed (Participants) | 76
Participants | 72

2. Primary Outcome: Number of Participants With AEs Leading to Study Drug Discontinuation
Description: Number of participants with AEs leading to study drug discontinuation was reported.
Time Frame: Up to 30 days after study treatment discontinuation (treatment exposure ranged from 1 to 82 months)
Population: OLAS included all data from participants who were enrolled into this open-label extension study, from the time they entered this open-label extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 Milligrams (mg)
Number analyzed (Participants) | 76
Participants | 9

3. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is any untoward medical occurrence that at any dose resulting in any of following outcomes: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product. Treatment-emergent SAEs were those events that started after administration of the first dose and up to safety follow-up visit/end of study, that is, 30 days after the last dose of study medication.
Time Frame: Up to 30 days after study treatment discontinuation (treatment exposure ranged from 1 to 82 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 Milligrams (mg)
Number analyzed (Participants) | 76
Participants | 44

4. Primary Outcome: Number of Participants With Hemoglobin Abnormalities
Description: Number of participants with hemoglobin abnormalities were reported. It included hemoglobin less than (<) 80 grams per liter (g/L), hemoglobin <100 g/L, hemoglobin greater than or equal to (>=) 80 g/L and <100 g/L, hemoglobin <100g/L and a decrease of >20 g/L from baseline, decrease of >20 g/L in hemoglobin from baseline, decrease of >20 g/L and <=50 g/L in hemoglobin from baseline, and decrease of >50 g/L in hemoglobin from baseline.
Time Frame: Up to 30 days after study treatment discontinuation (treatment exposure ranged from 1 to 82 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 Milligrams (mg)
Number analyzed (Participants) | 76
Participants
  Hemoglobin < 80 g/L | 0
  Hemoglobin <100 g/L | 7
  Hemoglobin >= 80 g/L and <100 g/L | 7
  Hemoglobin <100g/L and a decrease of >20 g/L from baseline | 6
  Decrease of >20 g/L in hemoglobin from baseline | 32
  Decrease of >20 g/L and <=50 g/L in hemoglobin from baseline | 31
  Decrease of >50 g/L in hemoglobin from baseline | 5

5. Primary Outcome: Number of Participants With Liver Tests Abnormalities
Description: Number of participants with liver tests abnormalities were reported. It included alanine aminotransferase (ALT) or aspartate aminotransferase (AST): >=3 x Upper limit of the normal range (ULN), >=3 and <5 x ULN, >=5 ULN, and >=5 and <8 x ULN, >= 8 x ULN, and total bilirubin >=2 x ULN.
Time Frame: Up to 30 days after study treatment discontinuation (treatment exposure ranged from 1 to 82 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 Milligrams (mg)
Number analyzed (Participants) | 76
Participants
  ALT or AST >=3 x ULN | 2
  ALT or AST >=3 and <5 x ULN | 1
  ALT or AST >=5 x ULN | 1
  ALT or AST >=5 and <8 x ULN | 0
  ALT or AST >=8 x ULN | 1
  Total Bilirubin >=2 x ULN | 8

6. Primary Outcome: Change From Baseline in Blood Pressure at Month 6
Description: Change from baseline in blood pressure at Month 6 (both systolic blood pressure [SBP] and diastolic blood pressure [DBP]) was reported.
Time Frame: Baseline and Month 6
Population: OLAS included all data from participants who were enrolled into this open-label extension study, from the time they entered this open-label extension study. Here, 'N' (number of participants analyzed) signifies participants evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Macitentan 10 Milligrams (mg)
Number analyzed (Participants) | 70
Millimeters of mercury (mmHg)
  SBP | -0.4 (13.15)
  DBP | -2.8 (9.51)

7. Primary Outcome: Change From Baseline in Pulse Rate at Month 6
Description: Change from baseline in pulse rate at Month 6 was reported.
Time Frame: Baseline and Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Macitentan 10 Milligrams (mg)
Number analyzed (Participants) | 70
Beats per minute | -1.1 (8.76)

8. Primary Outcome: Change From Baseline in Body Weight at Month 6
Description: Change from baseline in body weight at Month 6 was reported.
Time Frame: Baseline and Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Macitentan 10 Milligrams (mg)
Number analyzed (Participants) | 70
kilograms (kg) | -0.35 (2.871)

ADVERSE EVENTS:
Time Frame: Up to 30 days after study treatment discontinuation (treatment exposure ranged from 1 to 82 months)
Description: Open-label analysis set (OLAS) included all data from participants who were enrolled into this open-label extension study, from the time they entered this open-label extension study.
Arm/Group | Macitentan 10 Milligrams (mg)
All-Cause Mortality (participants affected / at risk) | 14/76
Serious Adverse Events (participants affected / at risk) | 44/76
Other Adverse Events (participants affected / at risk) | 67/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macitentan 10 Milligrams (mg) (N=76)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Angina Pectoris (Cardiac disorders) | 1 (1)
Aortic Valve Stenosis (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (3)
Atrial Flutter (Cardiac disorders) | 2 (2)
Atrial Tachycardia (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 4 (9)
Cardiac Failure Acute (Cardiac disorders) | 3 (3)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Right Ventricular Failure (Cardiac disorders) | 5 (8)
Arteriovenous Malformation (Congenital, familial and genetic disorders) | 1 (1)
Deafness Neurosensory (Ear and labyrinth disorders) | 1 (1)
Cataract (Eye disorders) | 1 (2)
Vision Blurred (Eye disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (2)
Gastric Polyps (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 1 (1)
Large Intestine Polyp (Gastrointestinal disorders) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1)
Peritoneal Adhesions (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 3 (3)
General Physical Health Deterioration (General disorders) | 2 (2)
Multiple Organ Dysfunction Syndrome (General disorders) | 1 (1)
Peripheral Swelling (General disorders) | 1 (2)
Pyrexia (General disorders) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Appendiceal Abscess (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Covid-19 Pneumonia (Infections and infestations) | 1 (1)
Neutropenic Sepsis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (5)
Pneumonia Parainfluenzae Viral (Infections and infestations) | 1 (1)
Pulmonary Tuberculosis (Infections and infestations) | 1 (1)
Pyelonephritis Acute (Infections and infestations) | 1 (1)
Pyelonephritis Chronic (Infections and infestations) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Septic Shock (Infections and infestations) | 2 (2)
Streptococcal Sepsis (Infections and infestations) | 1 (1)
Chemical Burns of Eye (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 3 (3)
Catheterisation Cardiac (Investigations) | 1 (1)
Chest X-Ray Abnormal (Investigations) | 1 (1)
Haemoglobin Decreased (Investigations) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diplegia (Nervous system disorders) | 1 (1)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pickwickian Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Angioplasty (Surgical and medical procedures) | 3 (10)
Arterial Angioplasty (Surgical and medical procedures) | 7 (23)
Pulmonary Endarterectomy (Surgical and medical procedures) | 1 (1)
Air Embolism (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Reperfusion Injury (Vascular disorders) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macitentan 10 Milligrams (mg) (N=76)
Anaemia (Blood and lymphatic system disorders) | 10 (11)
Cardiac Failure (Cardiac disorders) | 5 (5)
Cataract (Eye disorders) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 7 (11)
Oedema Peripheral (General disorders) | 11 (13)
Pyrexia (General disorders) | 4 (5)
Bronchitis (Infections and infestations) | 9 (14)
Covid-19 (Infections and infestations) | 6 (7)
Nasopharyngitis (Infections and infestations) | 9 (15)
Respiratory Tract Infection Viral (Infections and infestations) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 12 (21)
Urinary Tract Infection (Infections and infestations) | 7 (14)
Blood Bilirubin Increased (Investigations) | 5 (6)
Blood Creatinine Increased (Investigations) | 4 (4)
C-Reactive Protein Increased (Investigations) | 6 (6)
Haemoglobin Decreased (Investigations) | 13 (17)
Weight Decreased (Investigations) | 7 (8)
Hyperuricaemia (Metabolism and nutrition disorders) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (9)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 6 (6)
Dizziness (Nervous system disorders) | 8 (15)
Headache (Nervous system disorders) | 7 (10)
Syncope (Nervous system disorders) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 11 (12)

LIMITATIONS AND CAVEATS:
Study limitations included the open-label (OL), uncontrolled design, and small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Actelion for review at least 30 days prior to submission for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT02060721/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT02060721/SAP_001.pdf